CLINICAL TRIAL: NCT06624969
Title: Virtual Reality in Reducing Acute Orthopedic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Scott A. Helgeson, Consultant, Assistant Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-009261
Record Dates: First submitted 2024-09-17; First posted 2024-10-03 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Fractures
Keywords: pain control; orthopedic; fracture; hospital
MeSH Terms: conditions — Fractures, Bone; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Intervention with virtual reality
  Interventions: Other: virtual reality
- Standard of care (No Intervention): No virtual reality intervention

INTERVENTIONS:
Other: virtual reality — Virtual reality program to reduce pain in orthopedic fractures
  Arms: Virtual reality

SUMMARY:
The primary aim of this research is to show that a virtual reality (VR) service line is feasible and can sustain itself with the ability to take care of patients. Additionally, the investigators aim to learn about the limitations of a service line and provide a pathway for future improvements in building a VR service line that is optimally aligned with the user's needs. Secondary aims are to evaluate the clinical aspects of the patient's outcomes including length of stay, morphine equivalents in pain medicine required during the hospital stay, and user experiences.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with an orthopedic fracture
2. Able to participate fully in all aspects of the study
3. Able to understand and sign informed consent
4. Individuals with unaided vision or those who can correct their vision using contact lenses

   Exclusion Criteria:
5. Non-English speaking
6. Self-reported history of acute and/or chronic severe motion sickness
7. The presence of a facial/head deformity that will prohibit the wearing of a VR head mounted display.
8. Legally blind or deaf
9. Have had a seizure within the past 1 year
10. Have current (within the past 30 days) clinically significant acute or chronic progressive or unstable/uncontrolled neurologic disorder
11. Have a known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
opioid use | From date of enrollment which begins at hospital admission until the date of hospital discharge, assessed up to 5 weeks
  Change in opioid equivalents during hospital stay from hospital admission to discharge

SECONDARY OUTCOMES:
reduction in anxiolytics | From date of enrollment which begins at hospital admission until the date of hospital discharge, assessed up to 5 weeks
  Change in anxiolytics during the hospital admission from admission to discharge
hospital length of stay | From date of enrollment which begins at hospital admission until the date of hospital discharge, assessed up to 5 weeks
reduction in sleep aids prescribed | From date of enrollment which begins at hospital admission until the date of hospital discharge, assessed up to 5 weeks
  Change in sleep aids prescribed during the hospital stay from hospital admission to discharge
User experiences | obtained once on the day of hospital discharge, up to 5 weeks from study enrollment
  Subjective user experiences with the virtual reality program obtained at hospital discharge using a questionnaire with Likert scale answers showing higher scores to have better experiences with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Scott Helgeson, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No